CLINICAL TRIAL: NCT04064827
Title: A Phase 3, Prospective, Open-Label, Multicenter Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Paricalcitol Oral Solution for the Treatment of Secondary Hyperparathyroidism in Pediatric Subjects Ages 0 to 9 Years With Stage 5 Chronic Kidney Disease Receiving Peritoneal Dialysis or Hemodialysis
Brief Title: A Study to Evaluate Safety, Efficacy and Pharmacokinetics of Paricalcitol For Treatment of Secondary Hyperparathyroidism (SHPT) in Pediatric Participants With Stage 5 Chronic Kidney Disease (CKD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-617
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease (CKD); Secondary Hyperparathyroidism (SHPT)
Keywords: Chronic Kidney Disease; Paricalcitol; Hyperparathyroidism; Pediatric Subjects; Peritoneal Dialysis (PD); Hemodialysis (HD); Intact parathyroid hormone (iPTH)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Hyperparathyroidism | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants Receiving Paricalcitol (Experimental): Participants will be administered paricalcitol three times a week (TIW) but no more frequently than every other day for 24 weeks
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol oral solution (2.5 mcg/mL) will be administered with an oral dispenser

SUMMARY:
The main objective of this study is to evaluate the safety, efficacy and pharmacokinetics of paricalcitol oral solution in pediatric participants of ages 0 to 9 years with SHPT associated with stage 5 CKD receiving Peritoneal Dialysis (PD) or Hemodialysis (HD). The 24-week study is divided into two 12-week dosing periods (Dosing Period 1 followed by Dosing Period 2).

ELIGIBILITY:
Inclusion Criteria:

* Participant is currently diagnosed with and/or being treated for secondary hyperparathyroidism (SHPT).
* Participant must be diagnosed with chronic kidney disease (CKD) stage 5 receiving peritoneal dialysis (PD) or hemodialysis (HD) for at least 30 days prior to initial Screening.
* For entry into the Washout Period (for vitamin D receptor activator [VDRA] non-naive participants), the participant must meet the appropriate laboratory criteria based upon the participant's age as described in the protocol.
* For entry into the Dosing Period (for VDRA-naive participants or VDRA non-naive participants who have completed the Washout Period), the participant must meet the appropriate laboratory criteria based upon the participant's age as described in the protocol.

Exclusion Criteria:

* Participant is scheduled to receive a living donor kidney transplant within 3 months of Screening or is a kidney transplant recipient.
* Participant is expected to discontinue peritoneal dialysis (PD) or hemodialysis (HD) within 3 months of the initial Screening visit.
* Participant has had a parathyroidectomy within 12 weeks prior to Screening.
* Participant is taking maintenance calcitonin, bisphosphonates, glucocorticoids (in a dose equivalent to more than > 0.16 mg/kg/day or 5 mg prednisone/day, whichever is lower), 4 weeks prior to Dosing.
* Participant is receiving calcimimetics at the time of Screening or is expected to initiate calcimimetics at any time throughout the study.
* Participant is unable to take oral medications.

Ages: 0 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieve Positive Response During Dosing Period 1 | Up to Week 12
  Positive response is defined as having two consecutive >= 30% reductions from baseline in intact parathyroid hormone (iPTH) or two consecutive iPTH values in the target range between 150 picograms (pg)/milliliters (mL) to 300 pg/mL (16.5-33.0 picomole[pmol]/L).
Incidence of Hypercalcemia During Dosing Period 1 | Up to Week 12
  Incidence of hypercalcemia is defined as two consecutive, post-baseline, corrected calcium measurements above the normal participants's age-specific upper limit.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve a Positive Response During Dosing Period 2 | Week 12 through Week 24
  Positive response is defined as having two consecutive >= 30% reductions from baseline in iPTH or two consecutive iPTH values in the target range between 150 pg/mL to 300 pg/mL (16.5-33.0 picomole[pmol]/L).
Percentage of Participants Who Achieve a Positive Response During Dosing Periods 1 and 2 Combined | Up to Week 24
  Positive response is defined as having two consecutive >= 30% reductions from baseline in iPTH or two consecutive iPTH values in the target range between 150 pg/mL to 300 pg/mL (16.5-33.0 picomole[pmol]/L).
Percentage of Participants Who Achieve Two Consecutive >= 30% Reductions in iPTH From Baseline During Dosing Period 1 | Up to Week 12
  Participants who achieve two consecutive >= 30% reductions in iPTH will be evaluated.
Percentage of Participants Who Achieve Two Consecutive >= 30% Reductions in iPTH From Baseline During Dosing Period 2 | Week 12 through Week 24
  Participants who achieve two consecutive >= 30% reductions in iPTH will be evaluated.
Percentage of Participants Who Achieve Two Consecutive >= 30% Reductions in iPTH From Baseline During Dosing Periods 1 and 2 Combined | Up to Week 24
  Participants who achieve two consecutive >= 30% reductions in iPTH will be evaluated.
Percentage of Participants Who Achieve Two Consecutive iPTH Values Between 150 pg/mL to 300 pg/mL (16.5 - 33.0 pmol/L) During Dosing Period 1 | Up to Week 12
  Participants who achieve two consecutive iPTH values between 150 pg/mL to 300 pg/mL (16.5 - 33.0 pmol/L) will be evaluated.
Percentage of Participants Who Achieve Two Consecutive iPTH Values Between 150 pg/mL to 300 pg/mL (16.5 - 33.0 pmol/L) During Dosing Period 2 | Week 12 through Week 24
  Participants who achieve two consecutive iPTH values between 150 pg/mL to 300 pg/mL (16.5 - 33.0 pmol/L) will be evaluated.
Percentage of Participants Who Achieve Two Consecutive iPTH Values Between 150 pg/mL to 300 pg/mL (16.5 - 33.0 pmol/L) During Dosing Periods 1 and 2 Combined | Up to Week 24
  Participants who achieve two consecutive iPTH values between 150 pg/mL to 300 pg/mL (16.5 - 33.0 pmol/L) will be evaluated.
Incidence of Hypercalcemia During Dosing Period 2 | Week 12 through Week 24
  Incidence of hypercalcemia is defined as two consecutive, post-baseline, corrected calcium measurements above the normal participants's age-specific upper limit.
Incidence of Hypercalcemia During Dosing Periods 1 and 2 Combined | Up to Week 24
  Incidence of hypercalcemia is defined as two consecutive, post-baseline, corrected calcium measurements above the normal participants's age-specific upper limit.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- United States (14):
  - Arkansas Children's Hospital /ID# 225417, Little Rock, Arkansas
  - Stanford University School of Medicine - Redwood City /ID# 252150, Redwood City, California
  - Childrens National Medical Center /ID# 225991, Washington D.C., District of Columbia
  - Holtz Childrens Hospital, University of Miami /ID# 225636, Miami, Florida
  - Nicklaus Children's Hospital /ID# 210517, Miami, Florida
  - Emory University /ID# 140665, Atlanta, Georgia
  - Augusta University Medical Center /ID# 252149, Augusta, Georgia
  - Boston Children's Hospital /ID# 162863, Boston, Massachusetts
  - Duplicate_Levine Children's Specialty Center- Charlotte /ID# 216057, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 266045, Winston-Salem, North Carolina
  - Children's Hospital of Philadelphia - Main /ID# 213802, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center /ID# 210495, Dallas, Texas
  - University of Utah /ID# 140669, Salt Lake City, Utah
  - Seattle Children's Hospital /ID# 162861, Seattle, Washington
- School of Medicine University of Puerto Rico-Medical Science Campus /ID# 140663, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M11-617